CLINICAL TRIAL: NCT05044767
Title: Observational and Prospective Multicenter Study to Evaluate the Long-term (10 Years) Performance and Safety (10 Years) of ATF Implants and Lapé Médical Devices Implanted During Total Hip Arthroplasty or Hemiarthroplasty.
Brief Title: Study to Evaluate the Performance and Safety of ATF Implants and Lapé Médical Devices Implanted During Hip Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: ATF Implants (Industry)
Responsible Party: Sponsor
Other Study IDs: PEPS
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Arthroplasty, Hip, Replacement
MeSH Terms: interventions — Arthroplasty, Replacement, Hip; Hemiarthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: total hip arthroplasty — hip replacement surgery
  Other Names: hemiarthroplasty

SUMMARY:
Observational and prospective multicenter study to evaluate the long-term (10 years) performance and safety (10 years) of ATF Implants and Lapé Médical devices implanted during total hip arthroplasty or hemiarthroplasty.

DETAILED DESCRIPTION:
Observational and prospective multicenter study to evaluate the long-term (10 years) performance and safety (10 years) of ATF Implants and Lapé Médical devices implanted during total hip arthroplasty or hemiarthroplasty.

The post-market clinical follow-up study to be conducted by ATF Implants following this plan aims to collect data from the follow-up of patients before and after hip replacement surgery with implants manufactured by ATF Implants and Lapé médical. In current practice, the surgeon-investigator evaluates the patient pre- and post-operatively according to predefined criteria used in orthopedic surgery and more particularly in hp replacement surgery. Complications and adverse effects observed are also recorded.

The main objective is to gather clinical evidence to evaluate the survival rate of ATP Implants and Lapé médical hip prostheses over the long-term, namely 10 years.

The secondary objectives are to evaluate the performance and safety of the prostheses over the same period (i.e. 10 years), as well as to obtain feedback on the performance /intended use and safety of the surgical instruments required for implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Male or female indicated for hip replacement surgery with hip prosthesis manufactured by ATF Implants and/or Lapé médical;

There are different indications for hip replacement surgery. The main ones are listed below:

* Dysplasia
* Primary Coxarthrosis
* Secondary Coxarthrosis
* Perthes disease
* Epiphysiolysis
* Ankylosing spondylitis
* Trochanteric bursitis
* Arthritis
* Degenerative arthritis
* Post-traumatic arthritis
* Rheumatoid arthritis
* Femoral neck fracture
* Osteonecrosis
* Revision

Depending on the specificities of the devices (size, absence/presence of a coating, material), indications may vary. This information can be found in the instruction for use. It is the surgeon's responsibility to select the most appropriate prosthesis for a given patient according to the patient's medical records and the instruction for use in force at the time of the procedure accompanying the medical device.

Exclusion Criteria:

* There are various contraindications for hip arthroplasty. The main ones are listed below:

  * An acute or chronic, local or systemic infection
  * Severe muscular, neurological or vascular deficiency compromising the affected extremity
  * A bone defect or insufficient bone quality that may compromise the stability of the implant
  * Any concomitant disease (dysplastic coxarthrosis with extreme coxa valga, short neck and severe varus) that may affect the function of the implant
  * Sensitivity to the material (allergy) Depending on the specificities of the devices (size, absence/presence of a coating, material), contraindications may vary. This information can be found in the instruction for use of the devices.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female indicated for hip replacement surgery with hip prosthesis manufactured by ATF Implants and/or Lapé médical.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Long-term survival rate | 10 years
  Long-term survival rate of the prostheses (10 years) with failure defined as revision surgery when considering all causes using Kaplan-Meier method.

SECONDARY OUTCOMES:
hip joint function | before and after surgery (6 month, 2 years, 5 years, 7 years, 10 years)
  The evolution of hip joint function, and in this case the degree of physical disability before and after an intervention with Merle d'Aubigné score (PMA score) or Harris Hip Score (HHS score) or Parker score

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Laffargue, Pr, Principal Investigator — Clinique du Croisé Laroche
Locations (13):
- France (13):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Clinique des Cèdres, Cornebarrieu
  - Centre Ostéo-Articulaire des Cèdres, Échirolles
  - Hôpital privé Drôme Ardèche, Guilherand-Granges
  - Clinique du Croisé Laroche, Marcq-en-Barœul
  - Polyclinique Saint George, Nice
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - CHU de Poitiers, Poitiers
  - Clinique de l'Atlantique, Puilboreau
  - CHU St Etienne, Hôpital Nord, Saint-Etienne
  - Polyclinique Sainte Thérèse, Sète
  - Clinique de l'Orangerie, Strasbourg
  - Hôpital privé du Vert Galant, Tremblay-en-France